CLINICAL TRIAL: NCT03747380
Title: Pre-operative Inspiratory Muscle Training Program to Prevent Pulmonary Complications After Thoracic Surgery
Acronym: CT0076
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-7755
Record Dates: First submitted 2018-09-13; First posted 2018-11-20 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inspiratory muscle program (Experimental): Inspiratory muscle training preoperative with standard of care
  Interventions: Other: inspiratory muscle program
- no inspiratory muscle program (Other): standard of care: postoperative spirometry with enhanced recovery program in thoracic surgery
  Interventions: Other: inspiratory muscle program

INTERVENTIONS:
Other: inspiratory muscle program — pre-operative inspiratory muscular training program

SUMMARY:
Postoperative pulmonary complications are the most common complications after thoracic surgery. In the literature, pulmonary complications after thoracic surgery are present in more than 37.5% of patients. No study investigates the impact of preoperative inspiratory muscle exercises program on pulmonary complications after thoracic surgery.

DETAILED DESCRIPTION:
Postoperative pulmonary complications are the most common complications after thoracic surgery. In the literature, pulmonary complications after thoracic surgery are present in more than 37.5% of patients. Pulmonary complications include atelectasia, pneumonia and respiratory failure.

In order to reduce the pulmonary complications, other surgical specialties, such as cardiac and esophagus surgeries, use preoperative inspiratory muscle training programs. No study investigates the impact of preoperative inspiratory muscle exercises program on pulmonary complications after thoracic surgery.

Project Design:

Randomized study on patients at-risk of pulmonary complications. Two parallel groups are recruited for comparison between preoperative inspiratory muscle training program and the standard of care (without preoperative inspiratory muscle training program). In the study, 2 groups of 100 patients each are recruited in thoracic clinic. A recruitment period of approximately 8 months is needed in order to establish if the inspiratory muscular training significantly reduce the pulmonary complications in the patients at-risk. The P. value to determine a significant impact is 0.05 with a power of 0.80. We aim to reduce pulmonary complications with the inspiratory muscle training program by 50%.

Randomization Method:

Computerized, secure and anonymous randomization using a secure information program.

Population under study:

Recruitment in thoracic clinic, during the initial consultation for a thoracic surgery in the department of thoracic surgery of the University of Montreal Hospital Center, of a total of 200 patients. One hundred patients in the preoperative inspiratory muscle training group and 100 patients in the control group with usual care preoperatively (standard of care).

The study population is at-risk of pulmonary complications patients. The risk factors of pulmonary complications are patients over 70 years, presence of cough and sputum, diabetes, active smoking, FEV1 (forced expiratory volume per second) less than 75% or under respiratory pump, body mass index over 27 kg / m2, FEV1 less than 80%, Tiffeneau index less than 70%, NYHA II (New York Heart Association Classification) or sleep apnea.

Analysis A comparison of pulmonary complications after surgery in patients who participated in the inspiratory muscle training program and a control group who will have the usual care of a postoperative thoracic surgery.

After surgery, perioperative follow-up including perioperative complications, duration of hospitalization and complications and mortality after 30 days of surgery.

Satisfaction and motivation will be assessed postoperatively at discharge and at 30-day postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Pulmonary resection: segmental resection or lobectomy or bilobectomy
* With or without previous pulmonary resection
* Thoracotomy and minimally invasive surgery
* With or without neoadjuvant chemotherapy
* 1 or more risk factors for pulmonary complications (over 70 years, cough and sputum, diabetes, smoking, FEV1 less than 75% or under pump, BMI over 27 kg / m2, FEV1 less than 80%, TIFF less than 70%, NYHA II or sleep apnea)

Exclusion Criteria:

* Refusal of the patient
* Pregnancy
* Pneumonectomy
* FEV1 less than 30%
* DLCO less than 30%
* Vo2 MAX less than 10cc / min / kg
* Contraindication to respiratory physiotherapy - Myocardial infarction or cerebrovascular accident for less than 1 year, unstable angina, aneurysm, significant hemoptysis less than 90 days, muscular or neurological pathology constraining respiratory physiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 141 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Numbers of postoperative pulmonary complications | Up to 30 days after surgery

SECONDARY OUTCOMES:
Numbers of morbidity and mortality | Up to 30 days after surgery
Length of stay (by days) | Up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No